CLINICAL TRIAL: NCT07156617
Title: A Study on the Heterogeneity of Efficacy of Interventional Therapy Combined With Systemic Therapy for Liver Cancer Based on Multi-center Real-world Data
Status: Not yet recruiting | Type: Observational
Sponsor: Xuhua Duan (Other)
Responsible Party: Sponsor-Investigator, Xuhua Duan, The First Affiliated Hospital of Zhengzhou University, The First Affiliated Hospital of Zhengzhou University
Organization: The First Affiliated Hospital of Zhengzhou University (Other)
Other Study IDs: 2025-KY-1142-002
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: Hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Immunotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Interventional therapy combined with systemic therapy: Interventional therapy combined with systemic therapy is divided into three subgroups, including 1)DEB-TACE in Combination with Targeted Therapy；2） DEB-TACE in Combination with Targeted Therapy and Immunotherapy；3）DEB-TACE in Combination with Targeted Therapy, Immunotherapy, and Other Interventional Therapies.
  Interventions: Procedure: Interventional therapy; Drug: Systemic therapy

INTERVENTIONS:
Procedure: Interventional therapy — Interventional therapy
Drug: Systemic therapy — Targeted Therapy drugs include but are not limited to Lenvatinib, Apatinib, etc. Immunotherapy drugs include but are not limited to Camrelizumab, Tislelizumab
  Other Names: Targeted Therapy; Immunotherapy

SUMMARY:
The system assesses the heterogeneity of HCC patients in terms of therapeutic outcomes (such as rwPFS, ORR, PRO) and adverse reactions during the process of interventional therapy combined with systemic treatment. It explores the clinical characteristics and biomarker levels of patients related to heterogeneity and builds a machine learning model to predict the risk of adverse reactions, providing evidence support for the construction of a patient-centered individualized decision-making system.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥ 18 years old, gender not restricted; 2. Diagnosed with HCC through pathological or imaging examination, and meeting the diagnostic criteria of the "Primary Liver Cancer Diagnosis and Treatment Guidelines (2024 Edition)"; 3. Has received or plans to receive interventional therapy combined with systemic treatment (including but not limited to DEB-TACE combined with targeted therapy, DEB-TACE combined with targeted therapy and immunotherapy, DEB-TACE combined with targeted therapy and immunotherapy other local interventional treatments (such as HAIC, ablation, particle implantation, etc.)); 4. Has completed baseline clinical information and treatment records, can cooperate with the follow-up arrangement, and has the willingness and ability to complete the entire research process; 5. Signed the informed consent form.

Exclusion Criteria:

* 1. Diagnosed with liver metastatic cancer or other primary malignant tumors that are not HCC, or with concurrent other active primary malignant tumors; 2. Clearly have severe cognitive impairment, mental illness or confusion, and are unable to cooperate with the visit or fill out the scale; 3. Expected survival period is less than 3 months or clinical judgment indicates that follow-up cannot be completed; 4. Liver function is in decompensation, with Child-Pugh classification as C; 5. The investigator considers any other situation that is not suitable for participating in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hepatocellular carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
rwPFS | up to 2 years
  The definition of rwPFS is the time from the first administration of combined therapy to the first imaging assessment indicating tumor progression or death, whichever occurs first.

SECONDARY OUTCOMES:
ORR | up to 2 years
  ORR is defined as the proportion of patients who achieve complete remission (CR, Complete Response) and partial remission (PR, Partial Response) according to the mRECIST criteria.
rwOS | up to2years
  The rwOS is defined as the time from the first administration of combined therapy to the occurrence of any cause of death. If there is no death record for the patient, the last visit time will be used as the censored value.
rwTTP | up to2years
  The rwTTP is defined as the time from the first administration of combined therapy to the first imaging assessment revealing tumor progression.
PRO | up to2years
  The PRO score includes the scores of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) and its liver cancer module (EORTC QLQ-HCC18) that were filled out by the patients themselves.
AE | up to2years
  Adverse Event

CONTACTS AND LOCATIONS:
Locations (14):
- China (14):
  - The Second Affiliated Hospital of Hainan Medical Universsity, Haikou, Hainan
  - Xingtai No.5 Hospital, Xingtai, Hebei
  - Deng zhou People's Hospital, Dengzhou, Henan
  - The Second People's Hospital of Jiaozuo, Jiaozuo, Henan
  - Huai He Hospital of Henan University, Kaifeng, Henan
  - Luo Yang Central Hospital, Luoyang, Henan
  - The First Affiliated Hospital of Henan University of science and Technology, Luoyang, Henan
  - First People's Hospital of Shangqiu, Shangqiu, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Zhou Kou Central Hospital, Zhoukou, Henan
  - Wuxi No.5 People's Hospital, Wuxi, Jiangsu
  - Jiangxi Provincial People's Hospitail, Nanchang, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Second People's Hospital of Jiaozuo, Jiaozuo

IPD SHARING:
Plan to Share IPD: No